CLINICAL TRIAL: NCT07329504
Title: Effects of Aikido and Taijiquan Training on Joint Mobility, Reaction Time and Power Among Mixed Martial Arts Players
Brief Title: Effects of Aikido and Taijiquan Training Among Mixed Martial Arts Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0487
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Sports Physical Therapy
Keywords: Aikido Training; Taijiquan Training; Mixed Martial Arts Players

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aikido training (Experimental): This group will receive Aikido training to improve joint mobility, reaction time and power.
  Interventions: Other: Aikido training
- Taijiquan training (Experimental): This group will receive Taijiquan training tom improve joint mobility, reaction time and power.
  Interventions: Other: Taijiquan training

INTERVENTIONS:
Other: Aikido training — This group will receive Aikido training to improve joint mobility, reaction time and power.
  Arms: Aikido training
Other: Taijiquan training — This group will receive Taijiquan training tom improve joint mobility, reaction time and power.
  Arms: Taijiquan training

SUMMARY:
Mixed Martial Arts (MMA) is a physically demanding sport that requires athletes to maintain high levels of strength, flexibility, rapid response, and power. However, the intense focus on strength and endurance training in MMA can often result in neglecting joint health, flexibility, and relaxation techniques. Traditional martial arts, such as Aikido and Taijiquan, offer a complementary training approach emphasizing fluid movement, balance, and relaxation, which could be beneficial for MMA athletes. Aikido focuses on harmonizing movement and using an opponent's momentum to neutralize their power, while Taijiquan emphasizes controlled movements and internal power ("qi") to enhance body awareness and relaxation. This study investigates the effects of Aikido and Taijiquan on joint mobility, reaction time, and power among MMA athletes, aiming to determine whether these martial arts can enhance performance and reduce injury risk.

This randomized clinical trial will involve 17 MMA athletes divided into two groups: Group A (Aikido training) and Group B (Taijiquan training). Over an eight-week period, each group will engage in three weekly training sessions lasting 60-75 minutes. Key performance indicators, including joint mobility (Sit and Reach Test), reaction time (Catch the Ruler Test), and power (Vertical Jump Test), will be measured before and after the training program. Statistical analyses will be conducted using SPSS software, with significance set at p=0.05, employing the Wilcoxon signed-rank test and Mann-Whitney U test for within-group and between-group comparisons, respectively.

DETAILED DESCRIPTION:
It will be a Randomized Clinical Trial study.The sample size of the study will be 34 participants (19 in each group) through non probability sampling technique. Data will be collected from Pakistan sports board coaching center LHR & Roar Martial Arts Fitness Club Lahore.Data will be collected within 10 months after approval of synopsis.

Inclusion Criteria:

* Both male and female mixed martial arts players' age 18-30 years will be included.
* Participants must engage in physical activity (2-3 times a week) (20).
* Players have training experience of Aikido and Taijiquan training (21).
* Participants must have minimum one year experience of mixed martial arts training (22).

Exclusion Criteria:

* Participants with sustained injuries (fractures, sprains and stress) will be excluded.
* Pregnant and lactating females will be excluded.
* Those participants taking medicine will be excluded.
* Participants with known history of joint disease or chronic illness.
* Participants engaged in other high intensity physical training outside of MMA.

Data Collection Tools:

* Hip Joint mobility will be assessed using sit-to-reach test
* Reaction time will be evaluated through hexagon test.
* Power will be evaluated through vertical jump test

ELIGIBILITY:
Inclusion Criteria:

* Both male and female mixed martial arts players' age 18-30 years will be included.
* Participants must engage in physical activity (2-3 times a week) (20).
* Players have training experience of Aikido and Taijiquan training (21).
* Participants must have minimum one year experience of mixed martial arts training (22).

Exclusion Criteria:

* Participants with sustained injuries (fractures, sprains and stress) will be excluded.
* Pregnant and lactating females will be excluded.
* Those participants taking medicine will be excluded.
* Participants with known history of joint disease or chronic illness.
* Participants engaged in other high intensity physical training outside of MMA.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-11-02 (Actual)

PRIMARY OUTCOMES:
Sit to reach test | 8 weeks
  The Sit and reach test is one of the linear flexibility tests which helps to measure the extensibility of the hamstrings and lower back. The Sit and Reach Test measures lower back and hamstring flexibility, with normal scores varying by age and gender. For men, scores range from 24-34 cm 20-29 age and decrease slightly with age, while women score 27-36 cm in the same age range, also seeing a gradual decline over time. Higher scores indicate above-average flexibility, mid-range scores are average, and lower scores suggest limited flexibility
Hexagon test | 8 weeks
  The Hexagon Test is a simple, agility-based fitness assessment primarily used to evaluate an individual's quickness, balance, and coordination. It involves the participant standing at the center of a hexagon marked on the ground, typically with each side measuring about 24 inches. The participant must quickly jump over each line of the hexagon in a specific clockwise or counterclockwise sequence, aiming to complete three laps as fast as possible without stepping on the lines or losing rhythm
Vertical jump test | 8 weeks
  The Vertical Jump Test measures explosive leg power by assessing how high an individual can jump from a stationary position. The participant first records their standing reach height, then jumps as high as possible, with the height difference indicating the vertical jump score. High scores suggest strong leg power and athleticism, while lower scores indicate areas for improvement. For males, an "Excellent" jump is over 28 inches, "Above Average" is between 24-28 inches, "Average" is 20-24 inches, and "Below Average" is under 20 inches. For females, an "Excellent" score is over 24 inches, "Above Average" falls between 20-24 inches, "Average" is 16-20 inches, and "Below Average" is less than 16 inches

CONTACTS AND LOCATIONS:
Overall Officials: Iqra khan, MS-SPT, Principal Investigator — Riphah International University; Tasghir Nabi, MS-SPT, Principal Investigator — Riphah International University
Locations (1):
- Roar Martial Arts Fitness Club, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] James LP, Haff GG, Kelly VG, Beckman EM. Towards a Determination of the Physiological Characteristics Distinguishing Successful Mixed Martial Arts Athletes: A Systematic Review of Combat Sport Literature. Sports Med. 2016 Oct;46(10):1525-51. doi: 10.1007/s40279-016-0493-1. PMID 26993133
- [Background] Almasi T, Guey LT, Lukacs C, Csetneki K, Voko Z, Zelei T. Systematic literature review and meta-analysis on the epidemiology of methylmalonic acidemia (MMA) with a focus on MMA caused by methylmalonyl-CoA mutase (mut) deficiency. Orphanet J Rare Dis. 2019 Apr 25;14(1):84. doi: 10.1186/s13023-019-1063-z. PMID 31023387
- [Background] Bueno JCA, Faro H, Lenetsky S, Goncalves AF, Dias SBCD, Ribeiro ALB, da Silva BVC, Filho CAC, de Vasconcelos BM, Serrao JC, Andrade A, Souza-Junior TP, Claudino JG. Exploratory Systematic Review of Mixed Martial Arts: An Overview of Performance of Importance Factors with over 20,000 Athletes. Sports (Basel). 2022 May 24;10(6):80. doi: 10.3390/sports10060080. PMID 35736820
- [Background] van der Woude LHV, Houdijk HJP, Janssen TWJ, Seves B, Schelhaas R, Plaggenmarsch C, Mouton NLJ, Dekker R, van Keeken H, de Groot S, Vegter RJK. Rehabilitation: mobility, exercise & sports; a critical position stand on current and future research perspectives. Disabil Rehabil. 2021 Dec;43(24):3476-3491. doi: 10.1080/09638288.2020.1806365. Epub 2020 Aug 17. PMID 32805152
- [Background] Pimentel RE, Pieper NL, Clark WH, Franz JR. Muscle metabolic energy costs while modifying propulsive force generation during walking. Comput Methods Biomech Biomed Engin. 2021 Nov;24(14):1552-1565. doi: 10.1080/10255842.2021.1900134. Epub 2021 Mar 22. PMID 33749464